CLINICAL TRIAL: NCT01859624
Title: A Clinical Investigation of the Safety and Efficacy of Albuterol on Motor Function in Individuals With Late-onset Pompe Disease, Whether or Not Receiving Enzyme Replacement Therapy
Brief Title: Albuterol in Individuals With Late Onset Pompe Disease (LOPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00034177
Record Dates: First submitted 2013-05-08; First posted 2013-05-22 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Pompe Disease
Keywords: LOPD; Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albuterol (Experimental): This study includes the off-label administration of oral albuterol (4 mg pill) and tracking the effect of motor function at two additional visits, 6 and 12 weeks following the initiation of the study drug. The initial dose of albuterol will be a 4 mg daily for the first 6 weeks. If the 4 mg is well tolerated, the dose will be increased to 8 mg at the 6 week visit.
  Interventions: Drug: Albuterol

INTERVENTIONS:
Drug: Albuterol — Albuterol 4 mg

SUMMARY:
Albuterol is a drug approved by the US Food and Drug Administration (FDA) for treating breathing problems such as asthma. Studies have shown that albuterol may be beneficial in improving muscle function in people with late-onset Pompe disease. The purpose of this study is to evaluate whether albuterol is safe and effective for improving muscle function in people with late-onset Pompe disease, whether or not they are receiving enzyme replacement therapy (ERT). For this study, albuterol is considered an investigational drug. The word "investigational" means albuterol is not approved by the FDA for individuals with late-onset Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Pompe disease by blood acid alpha-glucosidase (GAA) assay and GAA gene sequencing
2. Age: 18+ years at enrollment

Exclusion Criteria:

1. Continuous invasive ventilation (via tracheostomy or endotracheal tube)
2. Clinically relevant illness within two weeks of enrollment including fever > 38.2o C, vomiting more than once in 24 hours, seizure, or other symptom deemed contraindicative to new therapy.
3. Chronic heart disease (Myocardial infarction, arrythmia, cardiomyopathy)
4. History of seizure disorder
5. Hypothyroidism
6. Pregnancy/Breast Feeding [Women of childbearing potential must have a negative urine pregnancy test at each study visit. In addition, at Screening/Baseline women of childbearing potential must have been using a medically acceptable contraceptive for at least 3 months prior to study enrollment OR the subject a) has a regular menstrual cycle, b) Day 1 (onset of menses) for the current cycle is known, and c) the urine pregnancy test can be administered within the first two weeks of the current cycle (between Days 1 and 14)]. The urine pregnancy test will be administered and interpreted by Stephanie Dearmey, Physician Assistant (PA-C), who has completed training from the Department of Obstetrics and Gynecology. Mrs. Dearmey will use a commercially available test kit specified by the point-of-care testing policies. If these criteria for urine pregnancy testing are not met at the Screening/Baseline visit, then a blood pregnancy test will be done.
7. Patients on a non-standard schedule for ERT; for example, weekly infusions as opposed to infusions every two weeks.

The use of the following concommitant meds is prohibited during the study:

* diuretics (water pill);
* digoxin (digitalis, Lanoxin);
* beta-blockers such as atenolol (Tenormin), metoprolol (Lopressor), and propranolol (Inderal);
* tricyclic antidepressants such as amitriptyline (Elavil, Etrafon), doxepin (Sinequan), imipramine (Janimine, Tofranil), and nortriptyline (Pamelor);
* Monoamine oxidase (MAO) inhibitors such as isocarboxazid (Marplan), phenelzine (Nardil), rasagiline (Azilect), selegiline (Eldepryl, Emsam), or tranylcypromine (Parnate); or
* other bronchodilators such as levalbuterol (Xopenex), bitolterol (Tornalate), pirbuterol (Maxair), terbutaline (Brethine, Bricanyl), salmeterol (Serevent), isoetherine (Bronkometer), metaproterenol (Alupent, Metaprel), or isoproterenol (Isuprel Mistometer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 24 weeks

SECONDARY OUTCOMES:
Change in forced vital capacity at 3 months | Baseline and week 12
Change in 6 minute walk test in 6 months. | Baseline and 24 weeks
  Assessed by physical therapist.

CONTACTS AND LOCATIONS:
Overall Officials: Dwight D Koeberl, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Koeberl DD, Li S, Dai J, Thurberg BL, Bali D, Kishnani PS. beta2 Agonists enhance the efficacy of simultaneous enzyme replacement therapy in murine Pompe disease. Mol Genet Metab. 2012 Feb;105(2):221-7. doi: 10.1016/j.ymgme.2011.11.005. Epub 2011 Nov 11. PMID 22154081
- [Result] Koeberl DD, Austin S, Case LE, Smith EC, Buckley AF, Young SP, Bali D, Kishnani PS. Adjunctive albuterol enhances the response to enzyme replacement therapy in late-onset Pompe disease. FASEB J. 2014 May;28(5):2171-6. doi: 10.1096/fj.13-241893. Epub 2014 Jan 17. PMID 24443373